CLINICAL TRIAL: NCT04173182
Title: Role of Peridiverticular and Colonic Mucosa Inflammation Based on Confocal Laser Endomicroscopy in the Prediction of Complicated Diverticular Disease
Brief Title: Confocal Laser Endomicrospy in Colonic Diverticular Disease
Status: Completed | Type: Observational
Sponsor: Instituto Ecuatoriano de Enfermedades Digestivas (Other)
Responsible Party: Principal Investigator, Carlos Robles-Medranda, Head of the Endoscopy Division, Instituto Ecuatoriano de Enfermedades Digestivas
Other Study IDs: PCLEDD
Record Dates: First submitted 2019-11-06; First posted 2019-11-21 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Diverticular Disease; Diverticulitis; Diverticula
Keywords: colonoscopy; diverticular disease
MeSH Terms: conditions — Diverticular Diseases; Diverticulitis; Diverticulum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Inflammation on pCLE: Patients with inflammatory findings in the peridiverticular and colonic mucosa (crypt fusion and distortion, bright epithelium, and dilated-prominent branching vessels)
  Interventions: Diagnostic Test: Probe-based confocal laser endomicroscopy evaluation
- No inflammation on pCLE: Patients with normal findings on pCLE evaluation of the peridiverticular and colonic mucosa (absence of inflammation)
  Interventions: Diagnostic Test: Probe-based confocal laser endomicroscopy evaluation

INTERVENTIONS:
Diagnostic Test: Probe-based confocal laser endomicroscopy evaluation — Colonoscopy with confocal laser endomicroscopy evaluation of the peridiverticular and colonic mucosa on patients with diverticular disease

SUMMARY:
Confocal laser endomicroscopy detects inflammatory markers undetectable during high definition endoscopy. The investigators aimed to evaluate the role of peridiverticular and colonic mucosa inflammation in the prediction of the complicated diverticular disease using confocal laser endomicroscopy evaluation in the peridiverticular area in consecutive patients.

DETAILED DESCRIPTION:
Diverticular disease of the colon is a prevalent condition in the western hemisphere. Currently there is an endoscopic classification system for classifying diverticular disease; however, white light endoscopic fails to accurately detect inflammation.

Confocal laser endomicroscopy offers a real-time, in-vivo evaluation of the colonic mucosa, with an adequate correlation to histological findings. The investigators aimed to evaluate the role of peridiverticular and colonic mucosa inflammation in the prediction of complicated diverticular disease.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years old
* Writeen informed consent provided.
* Endoscopic visualization of diverticular disease during colonoscopy.
* Adequate bowel preparation BBPS >2 in each colon segment

Exclusion Criteria:

* Under 18 years old.
* Refuse to sign written informed consent.
* Pregnancy or nursing.
* Previous colorectal surgery
* History of colorectal cancer
* Known allergy to fluorscein
* Uncontrolled coagulopathy
* History of complicated diverticular disease
* Patients with inflammatory bowel disease
* Patients with severe comorbidities: kidney and liver failure
* NSAIDs and antibiotics two weeks prior enrollment
* Historyh of alcohol or drug abuse
* Patients with severe mental illness
* Patients with incomplete evaluation of the colon

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with uncomplicated diverticular disease detected on colonoscopy and evaluation of peridiverticular and colonic mucosa assed via pCLE.
Sampling Method: Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
ocurrence of complicated diverticular disease | up to 12 months
  To predict the ocurrence of complications in colonic diverticular disease based on pCLE findings
ocurrence of complicated diverticular disease | up to 24 months
  To predict the ocurrence of complications in colonic diverticular disease based on pCLE findings

SECONDARY OUTCOMES:
peridiverticular and colonic mucosa inflammation based on pcle | index procedure
  • Presence of peridiverticular and colonic mucosa inflammation based on confocal laser endomicroscopy.
DICA classification | index procedure
  DICA classification system in all patients during initial colonoscopy.
ocurrence of complicated diverticular disease | 12 months and 24 months
  Ocurrence of complicated diverticular disease, assed up to 12 months after enrollment based on Hinchey Classification (III-IV).
ocurrence of surgical intervention | 12 months and 24 months
  • Ocurrence of surgical invertenvion for the management of complicated diverticular disease

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Robles-Medranda, Principal Investigator — Ecuadorian Institute of Digestive Diseases
Locations (1):
- Ecuadorian Institute of Digestive Diseases, Guayaquil, Guayas, Ecuador

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tursi A, Brandimarte G, Di Mario F, Andreoli A, Annunziata ML, Astegiano M, Bianco MA, Buri L, Cammarota G, Capezzuto E, Chilovi F, Cianci M, Conigliaro R, Del Favero G, Di Cesare L, Di Fonzo M, Elisei W, Faggiani R, Farroni F, Forti G, Germana B, Giorgetti GM, Giovannone M, Lecca PG, Loperfido S, Marmo R, Morucci P, Occhigrossi G, Penna A, Rossi AF, Spadaccini A, Zampaletta C, Zilli M, Zullo A, Scarpignato C, Picchio M. Development and validation of an endoscopic classification of diverticular disease of the colon: the DICA classification. Dig Dis. 2015;33(1):68-76. doi: 10.1159/000366039. Epub 2014 Dec 17. PMID 25531499
- [Background] Tursi A, Brandimarte G, di Mario F, Nardone G, Scarpignato C, Picchio M, Elisei W; DICA Italian Group. The "DICA" endoscopic classification for diverticular disease of the colon shows a significant interobserver agreement among community endoscopists. J Gastrointestin Liver Dis. 2019 Mar;28(1):23-27. doi: 10.15403/jgld.2014.1121.281.dic. PMID 30851168
- [Background] Tursi A, Elisei W, Picchio M, Nasi G, Mastromatteo AM, Di Mario F, Di Rosa E, Brandimarte MA, Brandimarte G. Impact of diverticular inflammation and complication assessment classification on the burden of medical therapies in preventing diverticular disease complications in Italy. Ann Transl Med. 2017 Aug;5(16):320. doi: 10.21037/atm.2017.06.39. PMID 28861417
- [Background] Tursi A, Brandimarte G, Di Mario F, Annunziata ML, Bafutto M, Bianco MA, Colucci R, Conigliaro R, Danese S, De Bastiani R, Elisei W, Escalante R, Faggiani R, Ferrini L, Forti G, Latella G, Graziani MG, Oliveira EC, Papa A, Penna A, Portincasa P, Soreide K, Spadaccini A, Usai P, Bonovas S, Scarpignato C, Picchio M; DICA Collaborative Group: Luigi Di Cesare; Lecca PG, Zampaletta C, Cassieri C, Damiani A, Desserud KF, Fiorella S, Landi R, Goni E, Lai MA, Pigo F, Rotondano G, Schiaccianoce G. Predictive value of the Diverticular Inflammation and Complication Assessment (DICA) endoscopic classification on the outcome of diverticular disease of the colon: An international study. United European Gastroenterol J. 2016 Aug;4(4):604-13. doi: 10.1177/2050640615617636. Epub 2015 Nov 13. PMID 27536372